CLINICAL TRIAL: NCT05120115
Title: Evaluating Optimal Weight Design Parameters of a Hip Exoskeleton Designed for Rehabilitation.
Brief Title: Optimization of Hip-exoskeleton Weight Attributes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001245; R01HD100416 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-11-15 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy; Gait, Frontal
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight distribution and placement (Experimental): Changing where weight is distributed on belt around pelvis, specifically, bilaterally, 4th lumbar area, unilaterally on the left side. Also changing amount of weight at 0, 4, 6 and 8 kg.
  Interventions: Other: Weight belt

INTERVENTIONS:
Other: Weight belt — Wearing belt around waist with various weights attached.

SUMMARY:
The investigators are examining how weight distribution affects the way people walk, in terms of joint kinematics, kinetics, and muscle activity. The investigators are measuring these quantities while people walk while wearing a weighted belt. The investigators distribute the weights and walk for specified periods. They hypothesize that greater weight will have a greater effect on walking.

DETAILED DESCRIPTION:
The purpose of this study is to examine how the amount and distribution of weight on the pelvis affects how people walk. The investigators two factors, weight and placement. They are examining how these factors affect muscle activation, joint motions and foot forces. The investigators plan to recruit 40 healthy adult individuals. Each of the 20 experimental conditions (3x3 factorial and one control condition with no weight) will be recorded immediately in a single session. The investigators hypothesize that weight amount, gait speed and weight distribution will all affect how people walk, which will lead towards optimized design of hip exoskeletons.

ELIGIBILITY:
Inclusion Criteria:

* Willing to commit to the full experimental session

Exclusion Criteria:

* Functionally relevant lower limb musculoskeletal injury

  * Functionally relevant osteoarthritis and weight bearing restrictions
  * Severe respiratory problems that restrict the wearer from using a metabolic rate apparatus
* Patients with cardiac issues may be included, but the cardiac issue will be noted in the health history questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- [Derived] Normand MA, Lee J, Su H, Sulzer JS. The effect of hip exoskeleton weight on kinematics, kinetics, and electromyography during human walking. J Biomech. 2023 May;152:111552. doi: 10.1016/j.jbiomech.2023.111552. Epub 2023 Mar 22. PMID 37004392

RESULTS

PARTICIPANT FLOW:
Groups:
- Weight and Placement: Changing weights on belt at 0, 4, 6 and 8 kg (weight factor) and lumbar, bilateral or unilateral placement on pelvis (placement factor)
Period: Overall Study
Arm/Group | Weight and Placement
Started | 21
no Weight | 21
4kg and Bilateral Weight Distribution | 21
6kg and Bilateral Weight Distriubtion | 21
8 kg and Bilateral Weight Distriubtion | 21
4 kg and Lumbar Weight Distriubtion | 21
6kg and Lumbar Weight Distriubtion | 21
8 kg and Lumbar Weight Distribution | 21
4kg and Unilateral Weight Distribution | 21
6kg and Unilateral Weight Distribution | 21
8kg and Unilateral Weight Distribution | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Healthy individuals
Groups:
- Weight and Placement: Changing where weight is distributed on belt around pelvis, specifically, bilaterally, 4th lumbar area, unilaterally on the left side. Also changing weight amounts at 4, 6 and 8 kg.
  Weight belt: Wearing belt around waist with various weights attached.
Arm/Group | Weight and Placement
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.7 (5.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
height [Mean (Standard Deviation); unit: cm] | 172 (7.58)
weight [Mean (Standard Deviation); unit: kg] | 65.9 (8.53)

OUTCOME MEASURES:

1. Primary Outcome: Pelvic Obliquity
Description: Amount of pelvic obliquity in response to weighted belt measured using optical motion capture
Time Frame: One day
Population: Healthy individuals
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Weight and Placement: Varying weight at 0, 4, 6 and 8 kg. Varying placement at bilateral, unilateral and lumbar areas of pelvis.
Arm/Group | Weight and Placement
Number analyzed (Participants) | 21
degrees
  No weight | -0.55 (2.79)
  4 kg and bilateral placement | -0.83 (2.89)
  6kg and unilateral weight distribution | -1.2 (3.05)
  8kg and unilateral weight distribution | -0.7 (2.97)
  4 kg and lumbar placement | -0.19 (2.91)
  6 kg and lumbar placement | 0.08 (2.93)
  8kg and lumbar weight distribution | 0.45 (2.94)
  4kg and unilateral | -0.76 (2.98)
  6kg and unilateral | -0.8 (2.83)
  8kg and unilateral | -1.15 (2.77)
Statistical Analysis 1: Comparison: Weight and Placement; Test type: Equivalence — Examined differences between conditions; p = 0.05, ANOVA — Used Tukey Honestly Significant Difference post-hoc test

2. Secondary Outcome: Knee Flexion Angle During Swing Phase
Description: Knee flexion angle range of motion measured using optical motion capture
Time Frame: One Day
Population: Healthy Individuals
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Weight and Placement
Number analyzed (Participants) | 21
degrees
  No weight | 68.8 (8.5)
  4 kg with bilateral | 67.66 (8.84)
  6 kg with bilateral | 68.03 (7.49)
  8 kg with bilateral | 67.99 (7.95)
  4 kg with lumbar | 66 (6.2)
  6kg with lumbar | 66.13 (7.01)
  8kg with lumbar | 67.4 (9.84)
  4kg with unilateral | 68.41 (8.09)
  6kg with unilateral | 68.02 (8.57)
  8kg with unilateral | 66.23 (6.72)
Statistical Analysis 1: Comparison: Weight and Placement; Test type: Equivalence — Differences between conditions; p = 0.05, Mixed Models Analysis — Used Tukey Honestly Significant Difference post-hoc test

3. Secondary Outcome: Integrated Gastrocnemius Muscle Activity During Preswing Phase of Walking
Description: EMG signals were normalized via the mean-dynamic method (Burden and Bartlett, 1999), centering the EMG signal around 1. For data analysis, the EMG signal was integrated along each gait phase to calculate the integrated EMG (iEMG) values. For the gastrocnemius, we extrated the iEMG during the pre-swing phase only. The iEMG was normalized to average during walking, resulting in arbitrary units.
Time Frame: One day
Population: Healthy Individuals
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Weight and Placement
Number analyzed (Participants) | 21
arbitrary units
  No weight | 1.16 (0.53)
  4 kg and bilateral | 1.14 (0.48)
  6kg and bilateral | 1.20 (0.55)
  8kg and bilateral | 1.23 (0.53)
  4kg and lumbar | 1.24 (0.66)
  6kg and lumbar | 1.20 (0.54)
  8kg and lumbar | 1.19 (0.56)
  4kg and unilateral | 1.19 (0.49)
  6kg and unilateral | 1.20 (0.51)
  8kg and unilateral | 1.10 (0.43)
Statistical Analysis 1: Comparison: Weight and Placement; Test type: Equivalence — Differences between conditions; p = 0.05, Mixed Models Analysis — Used Tukey Honestly Significant Difference post-hoc test

ADVERSE EVENTS:
Time Frame: 1 day
Description: No difference
Arm/Group | Weight and Placement
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT05120115/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT05120115/ICF_001.pdf